CLINICAL TRIAL: NCT05303636
Title: A Multicenter, Open-label, Controlled Study to Investigate the Effect of Either LF111 or Drospirenone Chewable Tablets on Bone Mineral Density in Adolescent and Adult Women in Comparison With Non-users of Hormonal Contraceptive Methods
Brief Title: LF111 or Drospirenone Chew vs Non-hormonal Contraceptive Methods on Bone Mineral Density in Adolescent and Adult Women
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Insud Pharma (Industry)
Collaborators: Chemo Research (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Factorial | Masking: None | Purpose: Screening
Other Study IDs: LF111/401; 2020-000412-30 (EudraCT Number)
Record Dates: First submitted 2022-03-22; First posted 2022-03-31 (Actual); Last update posted 2023-06-18 (Actual); Status verified 2023-02

CONDITIONS: Change in Bone Mineral Density; Bone Loss
Keywords: Osteoporosis
MeSH Terms: conditions — Bone Diseases, Metabolic; Osteoporosis | interventions — drospirenone; Tablets

STUDY DESIGN:
Intervention Model Description: Two cohorts: Cohort 1 (adolescents); Cohort 2 (adults)
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- Cohort 1 (adolescents aged 14-17) Hormonal Treatment Arm (Experimental): Subjects in the USA will choose to use the LF111 tablets or drospirenone (DRSP) 3.5 mg chewable tablets; 1/3 of subjects in the USA should receive DRSP 3.5 mg chewable tablets. Only LF111 will be available to subjects in Europe.
  Interventions: Drug: LF111 (drospirenone 4 mg oral tablet) or drospirenone (DRSP) 3.5 mg chewable tablet
- Cohort 1 (adolescents aged 14-17) Non-Hormonal Contraceptive Arm (No Intervention): Subjects in this group will not receive any investigational product. They will be free to use a non-hormonal contraceptive method of their choice. Non-hormonal contraceptive methods include barrier contraceptive methods (condoms, female condoms, cervical caps, diaphragms, and contraceptive sponges), double barrier methods, non-hormonal IUD (e.g., copper IUD), surgical female sterilization, vasectomized partner, spermicides, and sexual abstinence.
- Cohort 2 (adults aged 18-45) Hormonal Treatment Arm (Experimental): Subjects in the USA will choose to use the LF111 tablets or drospirenone (DRSP) 3.5 mg chewable tablets; 1/3 of subjects in the USA should receive DRSP 3.5 mg chewable tablets. Only LF111 will be available to subjects in Europe.
  Interventions: Drug: LF111 (drospirenone 4 mg oral tablet) or drospirenone (DRSP) 3.5 mg chewable tablet
- Cohort 2 (adults aged 18-45) Non-Hormonal Contraceptive Method Arm (No Intervention): Subjects in this group will not receive any investigational product. They will be free to use a non-hormonal contraceptive method of their choice. Non-hormonal contraceptive methods include barrier contraceptive methods (condoms, female condoms, cervical caps, diaphragms, and contraceptive sponges), double barrier methods, non-hormonal IUD (e.g., copper IUD), surgical female sterilization, vasectomized partner, spermicides, and sexual abstinence.

INTERVENTIONS:
Drug: LF111 (drospirenone 4 mg oral tablet) or drospirenone (DRSP) 3.5 mg chewable tablet — LF111 (drospirenone 4 mg tablet orally daily on days 1-24, followed by placebo tablet orally daily on days 25-28) or drospirenone (DRSP) 3.5 mg chewable tablet chewed daily on days 1-24, followed by placebo tablet chewed daily on days 25-28) (USA only). Subjects in the USA who choose to use the hormonal contraceptive method may choose between LF111 and DRSP 3.5 mg chewable tablets. The DRSP 3.5 mg chewable tablets are not available to subjects in Europe. Subjects in Europe who choose to use the hormonal contraceptive method will only receive LF111.
  Arms: Cohort 1 (adolescents aged 14-17) Hormonal Treatment Arm; Cohort 2 (adults aged 18-45) Hormonal Treatment Arm

SUMMARY:
The primary objective of this study is to evaluate the impact of LF111 and drospirenone (DRSP) 3.5 mg chewable tablets on bone mineral density (BMD) at the lumbar spine after 12 months (13 medication cycles) of investigation in comparison to non-hormonal contraceptive methods. Secondary objectives include further evaluating the impact of LF111 and DRSP 3.5 mg chewable tablets on BMD and bone turnover after 12 months (13 medication cycles) in comparison to non-hormonal contraceptive methods and assessing the general safety and tolerability of LF111 and DRSP 3.5 mg chewable tablets in comparison to non-hormonal contraceptive methods. Exploratory objectives include evaluating the impact of LF111 and DRSP 3.5 mg chewable tablets on body fat and lean mass after 12 months (13 medication cycles) of investigation.

DETAILED DESCRIPTION:
This is a Phase IV, prospective, multicenter, open-label, controlled, non-randomized trial in female subjects between 14 to 45 years of age who are postmenarcheal for at least two years and premenopausal. Subjects who choose to take the trial medication (LF111 tablet or drospirenone [DRSP] 3.5 mg chewable tablet [USA only]) will be compared to subjects who choose to use non-hormonal contraceptive methods, enrolled in a 1:1 ratio. Subjects will also be separated into two cohorts: cohort 1 as adolescents aged 14-17, and cohort 2 as adults aged 18-45.

At Visit 1 (screening), informed consent/assent will be obtained, and the screening procedures will be performed. At Visit 2 (allocation to treatment), after confirming the subject's eligibility, subjects who choose to use LF111 or DRSP 3.5 mg chewable tablets (USA only) for pregnancy prevention will be provided with LF111 or DRSP 3.5 mg chewable tablets. The subjects will attend additional on-site visits 6 months and 12 months after Visit 2 (end of investigational phase) or within one week after premature trial discontinuation for routine safety assessments.

The primary objective of this study is to evaluate the impact of LF111 and DRSP 3.5 mg chewable tablets on bone mineral density (BMD) at the lumbar spine after 12 months (13 medication cycles) of investigation in comparison to non-hormonal contraceptive methods. Secondary objectives include further evaluating the impact of LF111 and DRSP 3.5 mg chewable tablets on BMD and bone turnover after 12 months (13 medication cycles) in comparison to non-hormonal contraceptive methods and assessing the general safety and tolerability of LF111 and DRSP 3.5 mg chewable tablets in comparison to non-hormonal contraceptive methods. Exploratory objectives include evaluating the impact of LF111 and DRSP 3.5 mg chewable tablets on body fat and lean mass after 12 months (13 medication cycles) of investigation.

ELIGIBILITY:
Inclusion Criteria:

* Female subjects with regular menstrual cycles (postmenarcheal for at least two years and premenopausal) aged 14 to 45 years.
* Female subjects aged between 14 to 17 years (inclusive) will only be included provided that:

  * Applicable national, state, and local laws allow subjects in this age group to consent/assent to receive contraceptive services, and
  * All applicable laws and regulations regarding the informed consent/assent of the subjects to participate in clinical trials are observed.
* Systolic blood pressure < 140 mmHg, diastolic blood pressure < 90 mmHg at Visit 1, in sitting position after 5 minutes of rest.
* Menstruation restarted for at least 6 months since last pregnancy (only applicable for women that were pregnant).
* Be able and willing to provide written informed consent, or assent if the subject is an adolescent, prior to undergoing any trial-related procedures.
* Willing to use trial contraception for thirteen 28-day cycles (hormonal treatment arm) or to use non-hormonal contraceptive methods for the duration of the trial (non-hormonal contraceptive arm), respectively.

Exclusion Criteria:

* Contraindications to the use of LF111 or DRSP 3.5 mg chewable tablets (such as active arterial or venous thromboembolic disorders, liver tumors benign or malignant, hepatic impairment, renal impairment, adrenal insufficiency, presence or history of cervical cancer or progestin-sensitive cancers, known or suspected sex-steroid sensitive malignancies, undiagnosed abnormal uterine bleeding, undiagnosed vaginal bleeding, hypersensitivity to active substance or excipient) or adverse effects due to previous contraceptive use (for the hormonal treatment arm only).
* BMD Z-score below -1.50. The TBLH Z-score applies only to Cohort 1 (adolescents) and the total body Z-score applies only to Cohort 2 (adults) when assessing study eligibility.
* Low trauma fracture(s) defined as a fracture that results from a fall from a standing height or less, excluding fingers, toes, face, and skull.
* Medical conditions associated with low bone mass:

  * Metabolic bone disease such as osteogenesis imperfecta, Paget's disease of the bone, osteomalacia/rickets.
  * Collagen vascular diseases such as Marfan syndrome and Ehlers-Danlos syndrome.
  * Chronic kidney disease stage 3 with estimated glomerular filtration rate (eGFR) < 60 mL/min/1.73 m2 using the Bedside Schwartz equation for adolescents and the Modification of Diet in Renal Disease (MDRD) method for adult subjects.
  * Gastrointestinal (malabsorptive) disease including inflammatory bowel disease, gastric bypass surgery and current post-gastrectomy syndrome.
  * Liver disease.
  * Abnormal bone mineral metabolism (hypocalcemia/hypercalcemia, hypophosphatemia/hyperphosphatemia, hypomagnesemia).
* In adolescents only: Short stature defined as height-for-age percentile less than the fifth percentile.
* Use of progestin-only contraceptive pills in the previous month or use of implantable hormonal contraceptives in the previous 6 months.
* Laboratory values at screening which are considered clinically significant and which in the opinion of the investigator would be detrimental for participation in the study.
* Ongoing pregnancy or wish for pregnancy.
* Currently lactating or stopped lactating within the last 12 months.
* Eating disorders (e.g., anorexia nervosa, bulimia).
* Celiac disease.
* Endocrine disorders (e.g., diabetes, hypothyroidism or hyperthyroidism, hyperparathyroidism, Cushing's disease) not adequately controlled with a stable treatment regiment for > 2 months.
* Rheumatoid arthritis.
* Current or ever use of medications or supplements known to increase BMD including bisphosphonates, denosumab, teriparatide, abaloparatide, romosozumab, calcitonin, fluoride and strontium.
* Treatment with medications that are known to decrease bone mass:

  * Glucocorticoids (oral, intravenous, chronic inhaled, chronic extensive topical [> 3 months]) within the previous 3 months. Note: Subjects taking chronic oral/intravenous glucocorticoids (prednisone ≥ 2.5 mg daily for ≥ 3 months, or the equivalent) will have a washout period of 12 months.
  * Depo-medroxyprogesterone acetate within the previous 24 months (if duration of use was less than 2 consecutive years). Note: Subjects using depo-medroxyprogesterone acetate for a duration of use greater than 2 years will be excluded.
  * Aromatase inhibitors and/or raloxifene within the previous 24 months.
  * Anticonvulsants (phenytoin, phenobarbital, carbamazepine and valproate), anti-retroviral protease inhibitors, cyclosporine, heparin, warfarin, thiazolidinedione, SGLT-2 inhibitors, tricyclic antidepressants, chronic proton pump inhibitor (PPI) use (> 3 months), or selective serotonin reuptake inhibitors (SSRIs) within the previous 3 months.
* Conditions that preclude BMD measurement i.e. lumbar spine/bilateral hip surgery with hardware in place, abdominal clips, umbilical ring (not willing to remove) or weight that exceeds the DXA machine limitation.
* Any condition that, in the opinion of the investigator, may jeopardize the trial conduct according to the protocol.
* Persons committed to an institution by virtue of an order issued either by the judicial or other authorities.

Ages: 14 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 1710 (Estimated)
Dates: Start 2022-03-28 (Actual); Primary Completion 2026-07 (Estimated); Study Completion 2027-03 (Estimated)

PRIMARY OUTCOMES:
Cohort 1: Mean absolute change in lumbar spine (L1-L4) Z-score in adolescents | Baseline to 12 months
  Measured by dual-energy X-ray absorptiometry (DXA)
Cohort 2: Mean percentage change in lumbar spine (L1-L4) BMD in adults | Baseline to 12 months
  Measured by DXA

SECONDARY OUTCOMES:
Cohort 1: Mean absolute changes in lumbar spine (L1-L4) Z-score in adolescents (hormonal treatment arm only) | Baseline to 6 months
  Measured by DXA
Cohort 1: Mean absolute changes in Z-scores (femoral neck, total hip, and total body less head [TBLH]) in adolescents | Baseline to 6 months (hormonal treatment arm only) and to 12 months
  Measured by DXA
Cohort 1: Mean absolute and percentage changes in lumbar spine, femoral neck, total hip, and TBLH BMD in adolescents | Baseline to 6 months (hormonal treatment arm only) and to 12 months
  Measured by DXA
Cohort 1: Mean absolute and percentage changes in TBLH bone mineral content (BMC) in adolescents | Baseline to 6 months (hormonal treatment arm only) and to 12 months
  Measured by DXA
Cohort 1: Proportion of adolescent subjects with percentage changes in lumbar spine, femoral neck, total hip, and TBLH BMD by categories | Baseline to 12 months
  Categories are ≥ 0%, < 0% to -1.5%, < -1.5% to -3%, < -3% to -5%, < -5% to -8% and < -8%
Cohort 1: Proportion of adolescent subjects with absolute changes in Z-scores (lumbar spine, femoral neck, total hip, and TBLH) by categories | Baseline to 6 months (hormonal treatment arm only) and to 12 months
  Categories are ≥ 0.50, < 0.50 to 0.30, < 0.30 to 0, < 0 to -0.30, < -0.30 to -0.50 and < -0.50
Cohort 2: Mean absolute changes in lumbar spine (L1-L4) BMD in adults | Baseline to 12 months
  Measured by DXA
Cohort 2: Mean absolute and percentage changes in femoral neck, total hip, and total body BMD in adults | Baseline to 12 months
  Measured by DXA
Cohort 2: Mean absolute and percentage changes in BMD (lumbar spine, femoral neck, total hip, and total body) in adults (hormonal treatment arm only) | Baseline to 6 months
  Measured by DXA
Cohort 2: Proportion of adult subjects with percentage changes in lumbar spine, femoral neck, total hip, and total body BMD by categories | Baseline to 12 months
  Categories are ≥ 0%, < 0% to -1.5%, < -1.5% to -3%, < -3% to -5%, < -5% to -8% and < -8%
Cohort 2: Mean absolute changes in Z-scores (lumbar spine, femoral neck, total hip, and total body) in adults | Baseline to 6 months (hormonal treatment arm only) and to 12 months
  Measured by DXA
Cohort 2: Proportion of adult subjects with absolute changes in Z-scores (lumbar spine, femoral neck, total hip, and total body) by categories | Baseline to 6 months (hormonal treatment arm only) and to 12 months
  Categories are ≥ 0.5, < 0.5 to 0.3, < 0.3 to 0, < 0 to -0.3, < -0.3 to -0.5 and < -0.5
Changes in body weight and body mass index (BMI) | Baseline to 12 months
  Changes in body weight and body mass index (BMI)
Routine laboratory values | Baseline to 6 months and to 12 months
  Mean absolute and relative changes in routine laboratory values
Serum estradiol (E2) levels (hormonal treatment arm only) | Baseline to 6 months and to 12 months
  Mean absolute and relative changes in serum estradiol (E2) levels
Number of subjects with adverse events as a measure of safety | Up to 12 months following treatment
  Adverse events include laboratory and vital sign abnormalities that are considered clinically significant, require treatment, fulfill any serious adverse event criterion, or cause the subject to change the trial schedule and are judged by either the reporting investigator or the sponsor as having a reasonable causal relationship to the trial medication (drospirenone) or placebo comparator (non-hormonal contraceptive methods).

OTHER OUTCOMES:
Changes in body fat and lean mass | Baseline to 12 months
  Fat mass and lean mass will be expressed in grams (g). Changes will be summarized using descriptive statistics for baseline and percentage change from baseline by cohort and treatment group.

CONTACTS AND LOCATIONS:
Overall Officials: Enrico Colli, MD, Study Director — Chemo Research SL
Locations (20):
- United States (20):
  - Cactus Clinical Research, Inc., Phoenix, Arizona
  - Velocity Clinical Research, Denver, Colorado
  - Advanced Clinical Research Network, Coral Gables, Florida
  - Health Care Family Rehab & Research Center, Hialeah, Florida
  - Vital Pharma Research, Hialeah, Florida
  - Cornerstone Research Institute, Longwood, Florida
  - New Age Medical Research Corporation, Miami, Florida
  - Florida Pharmaceutical Research and Associates, Inc., South Miami, Florida
  - Comprehensive Clinical Research, LLC, West Palm Beach, Florida
  - M3 Wake Research, Inc., Sandy Springs, Georgia
  - Family Care Research, Boise, Idaho
  - Tandem Clinical Research, Marrero, Louisiana
  - Clinical Trials Management, LLC - Southshore, Metairie, Louisiana
  - Meridian Clinical Research, Norfolk, Nebraska
  - M3 Wake Research, Raleigh, North Carolina
  - Lillestol Research LLC, Fargo, North Dakota
  - Corpus Christi Women's Clinic, Corpus Christi, Texas
  - Signature Gyn Services, Fort Worth, Texas
  - TMC Life Research, Inc., Houston, Texas
  - Seattle Clinical Research Center, Seattle, Washington

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Rosenbaum P, Schmidt W, Helmerhorst FM, Wuttke W, Rossmanith W, Freundl F, Thomas K, Grillo M, Wolf A, Heithecker R. Inhibition of ovulation by a novel progestogen (drospirenone) alone or in combination with ethinylestradiol. Eur J Contracept Reprod Health Care. 2000 Mar;5(1):16-24. doi: 10.1080/13625180008500376. PMID 10836659
- [Background] Cibula D, Skrenkova J, Hill M, Stepan JJ. Low-dose estrogen combined oral contraceptives may negatively influence physiological bone mineral density acquisition during adolescence. Eur J Endocrinol. 2012 Jun;166(6):1003-11. doi: 10.1530/EJE-11-1047. Epub 2012 Mar 21. PMID 22436400
- [Background] Beksinska ME, Smit JA. Hormonal contraception and bone mineral density. Expert Rev of Obstet Gynecol. 2011;6(3);305-319.
- [Background] Weaver CM, Gordon CM, Janz KF, Kalkwarf HJ, Lappe JM, Lewis R, O'Karma M, Wallace TC, Zemel BS. The National Osteoporosis Foundation's position statement on peak bone mass development and lifestyle factors: a systematic review and implementation recommendations. Osteoporos Int. 2016 Apr;27(4):1281-1386. doi: 10.1007/s00198-015-3440-3. Epub 2016 Feb 8. PMID 26856587
- [Background] Rizzo ADCB, Goldberg TBL, Biason TP, Kurokawa CS, Silva CCD, Corrente JE, Nunes HRC. One-year adolescent bone mineral density and bone formation marker changes through the use or lack of use of combined hormonal contraceptives. J Pediatr (Rio J). 2019 Sep-Oct;95(5):567-574. doi: 10.1016/j.jped.2018.05.011. Epub 2018 Jun 28. PMID 29959901
- [Background] Schwartz GJ, Munoz A, Schneider MF, Mak RH, Kaskel F, Warady BA, Furth SL. New equations to estimate GFR in children with CKD. J Am Soc Nephrol. 2009 Mar;20(3):629-37. doi: 10.1681/ASN.2008030287. Epub 2009 Jan 21. PMID 19158356
- [Background] Pierce CB, Munoz A, Ng DK, Warady BA, Furth SL, Schwartz GJ. Age- and sex-dependent clinical equations to estimate glomerular filtration rates in children and young adults with chronic kidney disease. Kidney Int. 2021 Apr;99(4):948-956. doi: 10.1016/j.kint.2020.10.047. Epub 2020 Dec 8. PMID 33301749
- [Background] Carr B, Dmowski WP, O'Brien C, Jiang P, Burke J, Jimenez R, Garner E, Chwalisz K. Elagolix, an oral GnRH antagonist, versus subcutaneous depot medroxyprogesterone acetate for the treatment of endometriosis: effects on bone mineral density. Reprod Sci. 2014 Nov;21(11):1341-51. doi: 10.1177/1933719114549848. Epub 2014 Sep 23. PMID 25249568